CLINICAL TRIAL: NCT03737019
Title: How Does Education of Health Personnel With Acceptance and Commitment Therapy Affect the Extent of Medical Certificates of Sick Leave and Drug Prescriptions?
Brief Title: Effects of Acceptance and Commitment Therapy in Primary Health Care
Acronym: ACTPrimary
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Collaborators: County Councils of Region Östergötland, Kalmar and Jönköping (Unknown)
Responsible Party: Principal Investigator, Fredrik H Nystrom, MD PhD, consultant in internal medicine, professor of internal medicine, University Hospital, Linkoeping
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2018/323-32
Record Dates: First submitted 2018-10-30; First posted 2018-11-09 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Medical Certificates for Sick Leave and Drug Prescriptions
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Prospective non-randomized trial with one interventional group and a parallel group without intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT in County Council of Kalmar (Experimental): Group education with ACT in six primary health care centers in County Council of Kalmar
  Interventions: Behavioral: Education with Acceptance and Commitment Therapy
- Control health care centers of County Council of Jönköping (Placebo Comparator): Five primary health care centers of County Council of Jönköping that do not get education.
  Interventions: Other: Control, no intervention

INTERVENTIONS:
Behavioral: Education with Acceptance and Commitment Therapy — Group education with Acceptance and Commitment Therapy of the personnel at each center.
  Arms: ACT in County Council of Kalmar
Other: Control, no intervention — Control, no interventions.
  Arms: Control health care centers of County Council of Jönköping

SUMMARY:
How does education of health personnel with Acceptance and Commitment Therapy affect the extent of medical certificates of sick leave and drug prescriptions in primary health care centers in Kalmar compared with similar centers in Jönköping in which the personnel do not get such therapy?

DETAILED DESCRIPTION:
Five primary health care centers in the County Council of Jönköping who do not get education according to Acceptance and Commitment Therapy (ACT) serve as controls. Six primary health care centers in County Council of Kalmar, with the same total number of listed patients (about 45 000 in total per County Council) in their areas undergo group education according to ACT. Data on medical certificates of sick leave and drug prescriptions are taken from registries (this is routine in primary health care in Sweden) at baseline and after 6, 12 and 24 months in both regions. The personnel at both centers also fill out questionnaires about their own quality of life at baseline and after 12 months. The investigators also plan to interview about 20 subjects on these matters.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* working at the health care center

Exclusion Criteria:

* age less than 18 years
* do not work at the Health care center

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2020-10-05 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Extent of medical certificates of sick leave by the doctors | 24 months in total
  Data on entire extent of medical certificates, i.e. how many sick days that were certified by all doctors at the primary health care centers, for all patients treated, during the time period.
Prescription of drugs by the doctors | 24 months in total
  Data on all prescription of all different drugs, during the time period, made by all the doctors at the primary Health care centers that participate, to all patients that were treated.

SECONDARY OUTCOMES:
Assessment of how the education with ACT affect the personnel according to SF36 | 12 months
  Questionnaire SF36 is filled out by the personnel at baseline and after 12 months
Assessment of how the education with ACT affect the personnel according to KEDS | 12 months
  Questionnaire Karolinska Exhaustion Disorder Scale (KEDS) is filled out by the personnel at baseline and after 12 months
Assessment of how the education with ACT affect the personnel according to WAI | 12 months
  Questionnaire Work ability Index (WAI) is filled out by the personnel at baseline and after 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik H Nyström, MD, prof., Principal Investigator — Region Östergötland, Sweden; Fredrik Nyström, MD, Principal Investigator — Linkoeping University
Locations (2):
- Sweden (2):
  - Faculty of Medicine and Health Sciences, Linköping, Sverige
  - University Hospital of Linkoping, Linköping

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kadowaki A, Alvunger AK, Larsen HI, Persdotter A, Zak MS, Johansson P, Nystrom FH. Education of the primary health care staff based on acceptance and commitment therapy is associated with reduced sick leave in a prospective controlled trial. BMC Fam Pract. 2021 Sep 8;22(1):179. doi: 10.1186/s12875-021-01526-5. PMID 34496751